CLINICAL TRIAL: NCT07281131
Title: Testing the Impact of Pre-visit Priming as a Mechanism Across Multiple Medication Use Behavioral Targets in Primary Care Practice
Brief Title: Testing the Impact of Pre-visit Priming for Medications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Southern California (Other)
Responsible Party: Principal Investigator, Julie Lauffenburger, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2025P003030; 5P30AG024968 (NIH)
Record Dates: First submitted 2025-12-11; First posted 2025-12-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Deprescribing; Statin Prescribing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-visit patient prompts (Experimental): The intervention itself is a pre-visit prompt delivered prior to upcoming visits that includes a brief recommendation to the patient to discuss the medication use target with the PCP at the visit and a handout about the medication.
  Interventions: Behavioral: Pre-visit prompts
- Usual Care (No Intervention): No intervention delivery outside of regular clinical practice.

INTERVENTIONS:
Behavioral: Pre-visit prompts — The intervention itself is a pre-visit prompt delivered prior to upcoming visits that includes a brief recommendation to the patient to discuss the medication use target with the PCP at the visit and a handout about the medication. The medication targets include potentially-inappropriate medications and statin prescribing.
  Arms: Pre-visit patient prompts

SUMMARY:
We will use EHR data to identify eligible patients at BWH primary care clinics. Patients will be eligible if they have an upcoming primary care provider (PCP) appointment at an included BWH clinic, are ≥65 years, and are eligible for a medication target; exclusion criteria will include relevant EHR-documented allergies. After sharing patients with PCPs for potential opt-out, patients will be randomized 1:1 in REDCap® to intervention or usual care (no prompt). The intervention will include a pre-visit patient-facing prompt with information about the evidence-based medication target. If patients are eligible for multiple targets, one will be randomly selected. The primary clinical outcome will be measured on the day of the PCP visit using EHR data, depending on target: a) discontinuation or tapering order, or b) prescribing. Secondary outcomes will include a) these same measures in a 60-day follow-up period after the visit to capture any follow-up actions. We will use an intention-to-treat approach including patients regardless of whether the visit occurred. We plan to conduct the trial until 1700 patients are reached. We will also conduct exploratory mediation analyses of mechanisms through brief patient surveys with behavioral scales and PCP survey.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age
* Have an upcoming clinic appointment with a BWH PCP at one of the included clinics

In addition, they must meet the following eligibility criteria for at least one medication target behavior (based on EHR data):

1. Statin use for primary prevention (65-75 years of age): Having a EHR diagnosis or problem list documentation of: diabetes, hypertension, smoking, or high cholesterol and estimated eligible cardiovascular risk and no current outpatient prescription for a statin
2. High-risk medication use (≥65 years of age): Have an active outpatient prescription for ≥1 medication on the American Geriatrics Society Beers Criteria® List for Avoid Medications based on EHR records

Exclusion Criteria:

* Documented allergy to one of the components (statin).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Completion of medication prescribing/deprescribing target on day of PCP visit | 1 day
  The primary clinical outcome will be measured on the day of the primary care provider (PCP) visit through EHR data, depending on medication target: a) discontinuation or taper, or b) statin prescribing.

SECONDARY OUTCOMES:
Completion of medication prescribing/deprescribing target within 60 days | 60 days
  The secondary clinical outcome will be measured within the 60-day follow-up on or after the primary care provider (PCP) visit through EHR data, depending on medication target: a) discontinuation or taper, or b) statin prescribing.

IPD SHARING:
Plan to Share IPD: Yes
The project will result in a Limited Data Set and a de-identified data set of the outcomes, intervention arms, and sociodemographic and clinical characteristics.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: These data will be available upon request. To the extent the context of data collection can be revealed without compromising privacy and identity of research participants, it will be included. Algorithms and other programming code used to identify patients for the study and evaluate study outcomes will be available upon request. We will also provide the underlying logic to build the tools to other health systems upon request.
Access Criteria: Data will be controlled access with the General Research Use Data Use Limitation, as allowed by the informed consent and the institutional certification, anticipated through the Aging Research Biobank.